CLINICAL TRIAL: NCT05331300
Title: A Phase 1/2a, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Determine the Safety, Tolerability, Preliminary Efficacy, Immunogenicity and Pharmacokinetic Properties of LASN01 in Healthy Subjects and in Patients With Pulmonary Fibrosis or Thyroid Eye Disease
Brief Title: A Study to Evaluate the Safety, Preliminary Efficacy, and Pharmacokinetic Properties of LASN01 in Healthy Subjects and in Patients With Pulmonary Fibrosis or Thyroid Eye Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lassen Therapeutics 1 PTY LTD (Industry)
Responsible Party: Sponsor
Organization: Lassen Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: LASN01-CL-1101
Record Dates: First submitted 2022-03-16; First posted 2022-04-15 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Fibrosis; Thyroid Eye Disease
MeSH Terms: conditions — Pulmonary Fibrosis; Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- LASN01 - Parts A and B [Healthy Volunteers] (Experimental)
  Interventions: Drug: LASN01
- Placebo - Parts A and B [Healthy Volunteers] (Placebo Comparator)
  Interventions: Drug: Placebo
- LASN01 - Part C [Pulmonary Fibrosis] (Experimental)
  Interventions: Drug: LASN01
- Placebo - Part C [Pulmonary Fibrosis] (Placebo Comparator)
  Interventions: Drug: Placebo
- LASN01 - Part D [Thyroid Eye Disease] (Experimental)
  Interventions: Drug: LASN01
- Placebo - Part D [Thyroid Eye Disease] (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LASN01 — Escalating single and multiple doses of LASN01
  Arms: LASN01 - Parts A and B [Healthy Volunteers]
Drug: LASN01 — LASN01 will be administered intravenously
  Arms: LASN01 - Part C [Pulmonary Fibrosis]; LASN01 - Part D [Thyroid Eye Disease]
Drug: Placebo — Escalating doses of matching placebo
  Arms: Placebo - Parts A and B [Healthy Volunteers]
Drug: Placebo — Placebo will be administered intravenously
  Arms: Placebo - Part C [Pulmonary Fibrosis]; Placebo - Part D [Thyroid Eye Disease]

SUMMARY:
LASN01 is a novel, fully human antibody directed against the human IL-11 receptor that is being developed to address the fibro-inflammatory pathology of pulmonary fibrosis and TED. This study is a four-part trial consisting of Parts A, B, C and D.

The primary objective of this study is to evaluate the safety and tolerability of LASN01, and the secondary objective is to evaluate the preliminary efficacy, immunogenicity, and pharmacokinetics of single and multiple doses of LASN01 in healthy participants and in patients with idiopathic pulmonary fibrosis (IPF) or progressive fibrosing interstitial lung disease (PF-ILD) or Thyroid Eye disease (TED).

Please note that both the Phase 1 (single and multiple ascending dose, SAD/MAD) portion in healthy volunteers and the Phase 2a portion in patients are completed.

DETAILED DESCRIPTION:
This randomized, placebo-controlled clinical trial (LASN01-CL-1101) consists of 4 parts, each part containing adaptive design elements that can be modified.

In Phase 1, Part A comprised of a single-dose administration in healthy participants in 5 dose cohorts and Part B comprised of a multiple-dose administration in healthy participants in 2 dose cohorts. Parts A&B have been completed.

In the Phase 2a portion, Part C comprised of a multiple-dose administration in a single cohort of patients with IPF and PF-ILD, and Part D comprised of a multiple-dose design in a single cohort of patients with TED.

In each part of the study, participants were randomized to receive IV doses of LASN01 or placebo.

ELIGIBILITY:
I. Participant Inclusion Criteria-

Parts A, B, C, and D

1. Female participants must be nonpregnant, nonlactating, and either postmenopausal for ≥12 months, surgically sterile for ≥6 months, or agree to use 2 effective methods of contraception or a highly effective method of contraception. Males must be surgically sterile for ≥6 months or agree to highly effective methods of contraception.
2. Able to comprehend and willing to sign an ICF and understand and comply with the requirements of the study.

   Part A and Part B only
3. Males or females, 18 through 60 years of age, inclusive
4. Body weight ≥110 pounds (≥50 kg); body mass index (BMI) within the range of 18 through 32.0 kg/m2
5. In good health as determined by the Investigator

   Part C only
6. Male and female patients >40 years of age (IPF patients) or ≥21 years of age (PF-ILD patients)

   IPF-specific Inclusion Criteria:
7. A diagnosis of IPF
8. IPF has been stable for ≥3 months at Screening

   PF-ILD-specific Inclusion Criteria:
9. Patients with physician diagnosed ILD who fulfill ≥1 of the following criteria for PF-ILD within 24 months of the Screening visit despite treatment with approved and/or unapproved medications used in clinical practice to treat ILD.
10. Fibrosing lung disease on HRCT performed within 3 years of the Screening Visit
11. For patients with underlying CTD: stable CTD as defined by no initiation of new therapy or withdrawal of therapy for CTD within 6 weeks before the Screening visit
12. FVC ≥45% predicted

    Part D only
13. Male or female patients of age ≥18 years
14. Clinical diagnosis of Graves' disease associated with active TED
15. Moderate-to-severe active TED
16. Less than 15 months from onset of TED in the study eye
17. No previous medical treatment for TED with the exception of local supportive measures, mycophenolate and oral or injectable steroids, immunomodulating therapies, and/or orbital irradiation/radiotherapy

II. Participant Exclusion Criteria

Parts A, B, C, and D

1. Any acute or chronic condition that would limit the participant's ability to participate in and complete this clinical study

   Part A and Part B only
2. Significant history or clinical manifestation of any significant endocrine, metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
3. History of significant hypersensitivity; intolerance; or allergy to any drug compound, food, or other substance; or history of anaphylaxis or angioedema
4. Positive serum test for HIV or hepatitis infection
5. Currently receiving any antibiotics for upper or lower respiratory tract infections
6. Use of any prescription drug or vaccine within 21 days before Check-in with the exception of hormonal contraceptives and vaccines.
7. Any prescription biologic within 3 months or 5 half-lives (whichever is greater) before Check-in
8. Participation in any other investigational study drug trial in which an investigational study drug was administered within 30 days before randomization or an investigational biological study drug was administered within 3 months before Check-in

   Part C only
9. History of clinically relevant cardiovascular disease that could jeopardize a patient's health during the course of the study
10. Patients with concurrent active malignancy other than adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix

    IPF-specific Exclusion Criteria:
11. FVC <45% predicted of normal or a forced expiratory volume during the first second of the forced breath (FEV1)/FVC ratio of <0.7
12. Extent of emphysema in the lungs exceeds fibrosis
13. Currently receiving pirfenidone or nintedanib if on treatment for <3 consecutive months or needed dose modification due to AEs in the last 3 months

    PF-ILD-specific Exclusion Criteria:
14. Diagnosis of IPF
15. Diagnosis of sarcoidosis
16. Significant pulmonary arterial hypertension
17. FVC <45% predicted of normal or a FEV1/FVC ratio of <0.7
18. Previous treatment with pirfenidone

    Part D only
19. Any previous use of anti-insulin-like growth factor 1 receptor monoclonal antibody (eg, teprotumumab) at any time
20. Patients with 2 mm proptosis decrease between Screening and Baseline, or a 1-point decrease on the CAS 7-point scale in any 2 weeks during the Screening period
21. Patients with decreased best corrected visual acuity due to optic neuropathy, new visual field defect, or color defect secondary to optic nerve involvement within the last 6 months before Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Treatment emergent, treatment related, and serious adverse events | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1-Day 365 in Part D
Changes in concomitant medications | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1-Day 365 in Part D
Changes from Baseline in clinical laboratory evaluations following study drug administration | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1-Day 365 in Part D
Changes from Baseline in vital signs following study drug administration | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1-Day 365 in Part D
Changes from Baseline in 12-lead electrocardiogram (ECG) parameters following study drug administration | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1-Day 365 in Part D
Changes from Baseline in physical examination (PE) results following study drug administration | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1-Day 365 in Part D

SECONDARY OUTCOMES:
PK parameter assessed by serum LASN01 concentration at specified timepoints for maximum plasma concentration (Cmax) | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1- Day 365 in Part D
PK parameter assessed by serum LASN01 concentration at specified timepoints for time to peak concentration (T max) | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1- Day 365 in Part D
PK parameter assessed by serum LASN01 concentration at specified timepoints for area under curve (AUC) | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1- Day 365 in Part D
PK parameter assessed by serum LASN01 concentration at specified timepoints for clearance volume (CL) | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1- Day 365 in Part D
PK parameter assessed by serum LASN01 concentration at specified timepoints for terminal phase volume (Vz) | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1- Day 365 in Part D
PK parameter assessed by serum LASN01 concentration at specified timepoints for half life ( t1/2). | Day 1-Day 57 in Part A, Day 1-Day 71 in Part B, Day 1-Day 211 in Part C, Day 1- Day 365 in Part D
Percentage of patients with a ≥2 mm reduction from Baseline in proptosis in the study eye, (LASN01 versus placebo) without deterioration [≥2 mm increase] of proptosis in the fellow eye at Week 29 | Week 1-Week 29 in Part D
Mean change from baseline in proptosis of LASN01 patients versus placebo patients | Day 1- Day 365 in Part D

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Site AU05, Hurstville, New South Wales
  - Site AU03, Brisbane, Queensland
  - Site AU01, Melbourne, Victoria
- Site HK01, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No